CLINICAL TRIAL: NCT07399808
Title: CDK4/6 Inhibitors in Breast Cancer Elderly Patients: an Observational Ambispective Longitudinal Multicenter Study
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Angioletta Lasagna, Oncologist, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: BC_EP
Record Dates: First submitted 2025-11-17; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Old Age
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is one of the tumors with the highest incidence and current evidence indicates a higher prevalence in elderly patients (≥70 years) with a higher mortality rate due to immunosenescence, diagnostic delay and under treatment. Elderly patients are still poorly represented in clinical trials and the main indications for the treatment of the elderly population are extrapolated from the guidelines used in studies conducted predominantly on the younger population. In particular, these guidelines do not take into account the significant variability of elderly patients, in particular their comorbidities, performance status, physiological age and frailty.

The aim of this study is to improve understanding of the clinical efficacy and safety of CDK 4/6i in older women in a real-world setting compared to younger women.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* patients with solid tumours undergoing active systemic treatment with CDK4/6 for adjuvant disease

Exclusion Criteria:

* Patients who are unable to understand informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this cross-sectional study includes patients followed at the Medical Oncology Foundation IRCCS Policlinico San Matteo Pavia and Medical Oncology ICS Maugeri Pavia, suffering from solid tumors subjected to active systemic treatment with CDK4/6 for the disease in the adjuvant phase
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the toxicity rate (both hematological and non-hematological) of any severity level in elderly patients (≥70 years) during administration of CDK 4/6i. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  The primary objective of this study will be to evaluate the toxicity rate (both hematological and non-hematological) of any severity level in elderly patients (≥70 years) during CDK 4/6i administration. The primary endpoint will be the estimated incidence of toxicity (haematological and/or non-haematological) of any grade over a 12-month time window in elderly MBC and EBC patients (≥70 years) from our cohort of cancer patients treated with CDK 4/6i.

SECONDARY OUTCOMES:
Compare the toxicity rate between elderly and young MBC subjects; | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  The ratio of the toxicity rates (hematological and/or non hematological) of any degree over a time window of 12 months between elderly and younger EBC patients.
Compare the rate of switch therapies between elderly and younger EBC subjects; | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  the ratio of patients who switched therapy to the total number of treated patients.
Compare the rate of dose reductions between elderly and younger EBC subjects; | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  The ratio of patients who had a dose reduction to total number of treated patients.
Compare the invasive disease free survival (iDFS) between elderly and younger EBC subjects. | from the date of CDK 4/6i initiation to the date of first occurrence of ipsilateral invasive breast tumor recurrence, assessed up to 24 months
  The iDFS: calculated from the date of CDK 4/6i initiation to the date of first occurrence of ipsilateral invasive breast tumor recurrence, local/regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer, or second primary nonbreast invasive cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy